CLINICAL TRIAL: NCT03615287
Title: Assessment of Inflammation Load, Endothelial and Cardiac Function Before and After Medical and Surgical Treatment in Inflammatory Bowel Diseases
Brief Title: Assessing Cardiovascular Dysfunction Pre- & Post-treatment in Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor of Cardiology, University of Athens
Other Study IDs: 42/25-01-18
Record Dates: First submitted 2018-07-20; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Assessment of the inflammation load through analysis of the values of CRP, WBC, IL-6, TNFa
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 40 subjects undergoing Medical Treatment
- Group B: 40 subjects undergoing Surgical Treatment
- Group C: 40 control subjects

SUMMARY:
The aim of this study is to compare medical and surgery treatment in IBD patients and healthy controls, by assessing the endothelial and cardiac function and the inflammation status.

DETAILED DESCRIPTION:
The aim of this study is to compare medical and surgery treatment in IBD patients and healthy controls, by assessing the endothelial and cardiac function and the inflammation status.

In particular, three subject groups will be enrolled, as follows:

40 patients [Crohn's disease (CD) & ulcerative colitis (UC)] who will undergo medical treatment (Group A), 40 patients (CD & UC) who will undergo surgery (Group B) and a healthy control group (Group C) comprising 40 subjects.

Assessment of the inflammation load (CRP, WBC, IL-6, TNFa), the endothelial function (FMD, PWV, cIMT, endothelial glycocalyx) and the cardiac function - via echocardiographic parameters (systolic and diastolic echo values, tissue doppler imaging-GLS-strain rate) - will be carried out for every subject group in two phases: prior to treatment and four months after the treatment, as applicable.

The objective is to investigate whether there is a statistically significant reduction of endothelial and cardiac dysfunction following medical and surgery treatment in IBD patients as well as to examine associations across the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBD diagnosed > 6 months via biopsy confirming the diagnosis
* Patients with IBD at an advanced & non-controllable phase (IBD scores,clinical status, endoscopic and biochemical values) requiring the initiation of a new medical treatment or surgical intervention.

Exclusion Criteria:

* Coronary Artery Disease
* Peripheral Arterial Disease
* Thromboembolic Disease (acute or chronic)
* Heart failure of any cause
* Valvular Disease
* Congenital Heart Defect
* Heart Rhythm Disorder
* Stroke, Renal or liver failure, malignancy, endocrine disorder
* Other autoimmune disorder or angiitis
* IBD diagnosed < 6 months
* BMI > 40 Kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBD patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change of CFR | Just before treatment and four (4) months after treatment
  Change of coronary flow reserve values in echocardiography pre & post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Papaconstantinou, PhD, Study Chair — 2nd Department of Surgery Aretaieion Hospital-University of Athens-Greece
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece